CLINICAL TRIAL: NCT03397719
Title: Parent Feedback Intervention Study: A Randomized Controlled Trial
Brief Title: Parent Video Feedback Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1707018416
Record Dates: First submitted 2017-12-13; First posted 2018-01-12 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Autism Spectrum Disorder; Parent-Child Relations
Keywords: Autism Spectrum Disorder; Early Intervention; Parent-Mediated Intervention
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): This group will receive treatment as usual. Each participant will receive three hours of in-vivo parent coaching per week for 6 months.
  Interventions: Behavioral: Control Group
- Treatment Condition (Experimental): This group will receive an additional component which will involve videotaping parent/child interactions at home for thirty minutes a week. Each week, the therapist will select sections of the video to review with the parent during one of the parent coaching sessions.
  Interventions: Behavioral: Treatment Condition

INTERVENTIONS:
Behavioral: Treatment Condition — This group will receive three hours of parent coaching per week, one hour per week will involve feedback on parent usage of coached strategies based on parent recorded interactions with their children.
  Arms: Treatment Condition
Behavioral: Control Group — This group will receive in-vivo parent coaching three hours per week.
  Arms: Control Group

SUMMARY:
The purpose of this study is to use a randomized controlled trial to test the effectiveness of parent coaching sessions using video-based feedback, compared to the sessions without the use of video-based feedback on parent strategy use.

DETAILED DESCRIPTION:
This study is a randomized controlled trial of video-based feedback interventions for the parents of young children with autism spectrum disorder (ASD). In the beginning of the study, each participant will be randomized to the video-based feedback condition (treatment condition) or standard care procedure (control condition). All participants will be asked to implement the strategies taught during the sessions in the home environment (e.g., following the child's lead, sitting face-to-face). Participants randomized into the video-based feedback condition (treatment condition) will be asked to video-tape their interactions with their children (maximum 30 mins/week at home during free play, book reading, bath or meal time routines). The therapist then will review the tapes and then use the recorded sessions to give feedback on the parents' use of strategies in addition to providing in-vivo feedback based on the live interactions during the sessions. For parents whose children are randomized into the standard care condition, the families will receive coaching based on in-vivo sessions as described above. For all participants, a battery of assessment (diagnostic, developmental testing), will be administered at the beginning of the study participation, in the mid-point at 3 months, at the end of their 6-month participation of treatment sessions, and then at the follow-up period, 6 months after the end of their participation of the treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* All children who will be enrolled into the early intervention (EI) classroom at the Center for Autism and the Developing Brain (CADB) will be invited to participate in the study.

Exclusion Criteria:

* We do not have any exclusionary criteria as long as the children meet the inclusion criteria (families with children with ASD between 1-4 years who will be enrolling in the CADB early intervention classroom).

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Change in Brief Observation of Social Communication Change (BOSCC) | Baseline, months 1-6, and follow-up (12 months)
  This is a brief, play-based assessment that aims to measure short-term changes in social communication. Scores range from 0 to 60 with higher scores indicating more ASD symptoms.

SECONDARY OUTCOMES:
Change in Autism Diagnostic Observation Schedule-2 (ADOS-2) | Baseline, post (6 months), follow-up (12 months)
  This is a semi-structured play-based interaction that assesses for symptoms associated with an Autism Spectrum Disorder (ASD). Total calibrated severity score ranges from 0 to 10, with higher scores indicating more ASD symptoms.
Change in Beck Depression Inventory | Baseline, post (6 months)
  Self-report rating inventory that measures characteristic attitudes and symptoms of depression. Scores range from 0 to 63, with higher scores indicating higher degrees of depression.
Change in Beck Anxiety Inventory | Baseline, post (6 months)
  Self-report inventory used to assess anxiety levels in adults and adolescents. Scores range from 0 to 63, with higher scores indicating higher degrees of anxiety.
Change in Parent Stress Index | Baseline, post (6 months)
  Evaluate the magnitude of stress in the parent. Percentile scores range from 0 to 100, with higher scores indicating greater parenting stress.
Change in Behavior Rating Inventory of Executive Function-Preschool Version | Baseline, post (6 months)
  Standardized rating scale designed to specifically measure the range of behavioral manifestations of executive function in preschool-aged children

OTHER OUTCOMES:
Change in Parent Strategies Rating | Baseline, months 1-6, and follow-up (12 months)
  This is a rating scale that is currently under development. It will be used to rate the parents' utilization of the strategies they are being taught throughout the intervention.Scores range from 19 to 100. Higher scores indicate effective and appropriate use of strategies taught in NDBI.
Change in Mullen Scales of Early Learning (MSEL) | Baseline, post (6 months), follow-up (12 months)
  This is a structured cognitive assessment which measures a child's abilities in visual reception, fine motor, expressive language, and receptive language. It will be used to assess cognitive functioning. Early Learning Composite Score ranges from 49 to 155, with higher scores indicating higher developmental and cognitive functioning.
Change in Vineland Adaptive Behavior Scales, Third Edition (VABS-III) | Baseline, post (6 months), follow-up (12 months)
  This is a structured interview that a trained assessor administers to a parent in order to assess adaptive functioning across a variety of domains including communication, play and leisure, and social domains. Adaptive Behavior Composite Score ranges from 20 to 140, with higher scores indicating higher adaptive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: So Hyun Kim, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine Center for Autism and the Developing Brain, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are undecided.

REFERENCES:
- [Derived] Klein CB, Swain DM, Vibert B, Clark-Whitney E, Lemelman AR, Giordano JA, Winter J, Kim SH. Implementation of Video Feedback Within a Community Based Naturalistic Developmental Behavioral Intervention Program for Toddlers With ASD: Pilot Study. Front Psychiatry. 2021 Dec 2;12:763367. doi: 10.3389/fpsyt.2021.763367. eCollection 2021. PMID 34925094